CLINICAL TRIAL: NCT03682744
Title: Immunotherapy for Peritoneal Carcinomatosis (IPC) - A Phase I Study of the Safety and Efficacy of Anti-CEA CAR-T Cell Intraperitoneal Infusions for Treatment of CEA-Expressing Adenocarcinoma Peritoneal Metastases or Malignant Ascites
Brief Title: CAR-T Intraperitoneal Infusions for CEA-Expressing Adenocarcinoma Peritoneal Metastases or Malignant Ascites (IPC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 340-74
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Peritoneal Carcinomatosis; Peritoneal Metastases; Colorectal Cancer; Gastric Cancer; Breast Cancer; Pancreas Cancer; Carcinoembryonic Antigen
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Breast Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anti-CEA CAR-T cells (Experimental): One intraperitoneal infusion of gene-modified anti-CEA T cells are administered to patients with CEA-expressing peritoneal metastases or malignant ascites
  Interventions: Biological: anti-CEA CAR-T cells

INTERVENTIONS:
Biological: anti-CEA CAR-T cells — Intraperitoneal delivery of anti-CEA CAR-T cells
  Other Names: Gene modified patient T cells; Designer T cells

SUMMARY:
This is an open-label, dose-escalation, phase I trial of the safety and efficacy of anti-CEA intraperitoneal CAR-T infusions for treatment in patients with CEA-expressing adenocarcinoma peritoneal metastases or malignant ascites.

DETAILED DESCRIPTION:
Patients undergo leukapheresis from which peripheral blood mononuclear cells are purified. T cells are activated and then re-engineered to express chimeric antigen receptors (CARs) specific for CEA. Cells are expanded in culture and returned to the patient by intraperitoneal infusion at specific cell doses. One anti-CEA CAR-T dose per patient is planned. Additional cycles may be administered at the discretion of the principal investigator. Normal peritoneal and tumor biopsies will be obtained at the time of the CAR-T infusion, on the final day of the treatment period, and during reporting interval #3.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Must have documented CEA+ carcinomatosis or malignant ascites as demonstrated by an elevated serum CEA level (≥ 10 ng/mL) or immunohistochemistry on a biopsy or cytologic specimen (archived tissue is acceptable), for determination of CEA expression. Primary tumor may be intact and limited liver and/or lung disease permitted.
3. Must have at least evaluable disease by physical examination, serum tumor markers, radiologic assessment, tumor markers, or laparoscopic visual assessment.
4. Have a life-expectancy ≥ 12 weeks and ECOG performance status ≤ 2.
5. May have low volume of liver metastases defined as < 50% replacement of the liver volume by metastatic disease, as long as all other eligibility criteria are satisfied.
6. Be willing and able to comply with the study schedule and all other protocol requirements.

Exclusion Criteria:

1. Female patients of childbearing age will be tested for pregnancy. Pregnant patients will be excluded from the study. Males who are actively seeking to have children will be made aware of the unknown risks of this study protocol on human sperm and the need to practice birth control.
2. Received an investigational study drug within 14 days of leukapheresis or 28 days before receiving first dose of study drug. Exceptions may be granted with medical monitor approval.
3. Received any approved anticancer medication within 14 days of leukapheresis or 14 days before receiving the first dose of study drug. Exceptions may be granted with medical monitor approval.
4. Have any unresolved toxicity > Grade 2 from previous anticancer therapy, except for stable chronic toxicities (≤ Grade 3) that are not expected to resolve.
5. Have a history of histologically confirmed metastases outside the peritoneal cavity, lungs, or liver.
6. Have high volume lung or liver metastases, defined as >5 lung lesions greater than 1 cm in size or ≥ 50% replacement the liver volume by metastatic disease.
7. Received CAR-T, CAR-T cell line, CAR-NK, CAR-pNK, or CAR-NK cell line therapies.
8. Have any of the following laboratory results at Screening (Screening volumes must be independent of blood product treatment):

   1. Hemoglobin ≤ 8.0 g/dL
   2. Platelet count < 50 × 109/L
   3. Absolute neutrophil count (ANC) < 1.0 × 109/L
9. Untreated or ongoing intra-abdominal infection or bowel obstruction.
10. Have any of the following laboratory results at Screening, regardless of causality:

    1. Serum creatinine ≥ 3.0, or estimated creatinine clearance ≤ 30 mL/min and not dialysis dependent
    2. Aspartate aminotransferase (AST) ≥ 4 × upper limit of normal (ULN) and total bilirubin ≥ 2.0 mg/dL (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).
11. Have human immunodeficiency virus (HIV) infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia, or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being HBsAg positive, or anti-HBc-antibody positive), or are positive for HBV deoxyribonucleic acid (DNA). HCV ribonucleic acid (RNA) must be undetectable by laboratory test.
12. Are pregnant or breastfeeding.
13. Have active bacterial, viral, or fungal infection: patients with ongoing use of prophylactic antibiotics, antiviral agents, or antifungal agents remain eligible as long as there is no evidence of active infection.
14. Has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
15. Has any condition, including the presence of laboratory abnormalities that places the patient at an unacceptable risk if the patient was to participate in the study.
16. Left ventricular ejection fraction (LVEF) < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Safety of Intraperitoneal CAR-T Cell Infusions as Measured by Number of Participants with Adverse Events | 16 weeks
  To determine the safety and maximum tolerated dose (MTD) following intraperitoneal infusion(s) of anti-CEA CAR-T cells for inoperable CEA+ peritoneal metastases or malignant ascites.

SECONDARY OUTCOMES:
Progression-Free Survival | 20 weeks
  As a measure of activity, Progression-free survival (PFS) will be assessed. The events for the assessment of PFS are disease progression and death events
Overall Survival | 20 weeks
  As a measure of activity, Overall Survival (OS) will be assessed. The events for the assessment of OS are death events.
Bowel Obstruction Free Survival | 20 weeks
  Measuring the time frame in which a patient does not experience a bowel obstruction
Changes in Quality of Life | 20 weeks
  Changes in quality of life measured by Quality of Life Index (IQI) survey pre and post-treatment
Response by the Peritoneal Carcinomatosis Index (PCI) | 16 weeks
  Direct visualization of tumor burden assessment by the PCI pre and post-treatment
Radiographic treatment response by MRI | 20 weeks
  Changes in tumor size
Radiographic treatment response by PET | 20 weeks
  Changes in tumor metabolic activity
Serologic response rates | 20 weeks
  Measurement of CEA and CA19-9

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Katz, MD, Principal Investigator — Roger Williams Medical Center
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roger Williams Medical Center, Providence, Rhode Island